CLINICAL TRIAL: NCT04404894
Title: Long-Term Prospective Registry to Evaluate Treatment Decisions and Clinical Outcomes in Prostate Cancer Patients From Diverse Urology Practice Settings Following Prolaris® Testing
Brief Title: Long-Term Prospective Registry in Prostate Cancer Patients From Diverse Urology Practice Settings Following Prolaris® Testing
Status: Active, not recruiting | Type: Observational
Sponsor: Myriad Genetic Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: URO-013
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Active Surveillance; Active Surveillance Durability; Prostate Cancer Treatment Selection; Prostate Cancer Risk Stratification; Prostate Cancer Oncological Outcomes
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prolaris tested patients with Prostate Cancer: Recently diagnosed patients with histologically proven, localized adenocarcinoma of prostate determined via transrectal ultrasonography and biopsy of at least 10 prostate sites who have undergone Prolaris testing.

SUMMARY:
This registry will evaluate treatment selection for patients with newly diagnosed, localized prostate cancer following Prolaris testing. It will measure the proportion of men who initially select treatment with active surveillance, the time frame between active surveillance selection and any change in treatment, and clinical outcomes.

DETAILED DESCRIPTION:
To evaluate use of the Prolaris score in treatment management decisions in an ethnically and racially diverse population of men who have been newly diagnosed with prostate cancer and who are potential candidates for active surveillance. This registry will evaluate oncologic and co-morbidity outcomes in patients who receive Prolaris testing. Additionally, the registry will measure the prevalence and distribution of pathogenic mutations in hereditary cancer risk-associated genes among men with prostate cancer who meet National Cancer Center Network (NCCN) criteria for hereditary cancer genetic testing.

The primary objective of this registry is to evaluate initial selection of active surveillance (Active Surveillance selection) versus definitive therapy (DT) among men with newly diagnosed prostate cancer who make treatment decisions with Prolaris testing, and among patient subsets defined by race/ethnicity.

The secondary objectives of the registry are to evaluate progression of from Active Surveillance to definitive therapy over time and prostate cancer-associated morbidities that affect quality of life among men with newly diagnosed prostate cancer and who undergo Prolaris testing, and among patient subsets defined by racial/ethnic background and ancestry.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older on date of enrollment.
* Diagnosed within the past six months with histologically proven, localized adenocarcinoma of prostate determined via transrectal ultrasonography and biopsy of at least 10 prostate sites.
* Received Prolaris testing and a resulting CCR score from the diagnostic biopsy sample as standard of care.
* Can be monitored for disease progression according to standard of care (e.g., current NCCN guidelines).

Exclusion Criteria:

* Estimated life expectancy < 10 years.
* Clinical evidence of metastasis or lymph node involvement.
* Received pelvic radiation prior to biopsy.
* Received androgen deprivation therapy (ADT) prior to biopsy; however, 5 alpha- reductase inhibitor (5-ARI) use is permitted.
* Plan to use PrCa-specific prognostic testing other than PSA for treatment decision making during Active Surveillance.
* Currently participating in an interventional clinical trial.
* Unable to provide routine clinical informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Urology Practices
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Active Surveillance (AS) selection versus Definitive Therapy (DT | 1 Year
  The primary endpoint of the registry is Active Surveillance selection, defined as the proportion of all men who select Active Surveillance in lieu of definitive therapy following confirmatory diagnosis of localized Prostate Cancer and Prolaris testing. Active Surveillance selection is
  documented by the treating provider and reflects the patient-provider decision at the time to pursue Active Surveillance with no curative intent.

SECONDARY OUTCOMES:
Active Surveillance Durability; Comorbidities | Active Surveillance durability, date of diagnostic biopsy will be recorded as the Active Surveillance initiation date. Definitive treatments collected at baseline and annually up to 10 years Comorbidities collected annually up to 10 years.
  Active Surveillance durability, measured as the length of time between the Active Surveillance initiation date and the first definitive therapy date. Comorbidities, including voiding problems, erectile dysfunction, bowel dysfunction, stress or urgency incontinence, depression, and anxiety, as measured by validated, standard of care quality-of-life assessments: the Expanded Prostate Cancer Index Composite Instrument (EPIC-26) and the Generalized Anxiety Disorder scale (GAD-7).

OTHER OUTCOMES:
Disease Progression | Baseline to year 10
  • Disease progression, measured as the proportion of men who:
  * Initiate and remain on Active Surveillance and subsequently experience distant metastasis or disease-specific mortality.
  * Initiate Active Surveillance and proceed to definitive therapy, or initially select definitive therapy, and subsequently experience biochemical recurrence (BCR), distant metastasis or disease-specific mortality. For radical prostatectomy (RP) patients, BCR is defined as PSA >0.2 ng/mL on at least two occasions more than two weeks apart or initiation of any salvage therapy greater than or equal to 6 months after surgery. For patients treated by external beam radiation therapy (EBRT), BCR is defined by reaching a post-EBRT PSA of nadir + 2 ng/mL (Phoenix criteria) or initiation of any salvage therapy 6 months after radiation.
Disease reclassification | Baseline to year 10
  Disease reclassification, defined as a patient initially treated with Active Surveillance for whom follow-up biopsy results in reclassification of the disease into a different NCCN risk category.
Baseline Clinicopathologic measures | Baseline to year 10
  Baseline clinicopathologic measures, including pre-biopsy PSA, date of biopsy, prostate volume, biopsy findings, total number of biopsy cores, number of positive cores, clinical stage, Gleason score, NCCN risk category, and Prostate Magnetic Resonance Imaging (MRI) assessment results with Prostate Imaging Reporting and Data System (PI-RADS) score(s) when available.
The Proportion of Men with PrCa who: | Baseline to year 10
  (1) Meet NCCN hereditary high-risk criteria, (2) undergo and complete hereditary cancer genetic testing; and (3) are found to carry pathogenic variants in tested cancer-predisposition genes.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Rayford, M.D., Principal Investigator — The Urology Group
Locations (7):
- United States (7):
  - Urology Centers of Alabama, Homewood, Alabama
  - VA Long Beach Healthcare System, Long Beach, California
  - Manatee Medical Research Institute, Bradenton, Florida
  - UroPartners, LLC, Westchester, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - The Urology Group, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No